CLINICAL TRIAL: NCT01473615
Title: Mindfulness Based Cognitive Therapy for Chronic Pain and Comorbid Unipolar Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Heidi Ashih, Principal Investigator, Clinical Instructor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011P001699
Record Dates: First submitted 2011-11-09; First posted 2011-11-17 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Major Depressive Disorder; Dysthymic Disorder; Depressive Disorder NOS; Chronic Pain
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder; Depression; Chronic Pain | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment As Usual + Mindfulness Based Cognitive Therapy (Experimental): Subjects randomized into the intervention group will receive, a manualized 8-week MBCT group skills program with sessions that each last 2 hours, in addition to their treatment as usual (TAU).
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy
- Treatment As Usual (No Intervention): Patients randomized into the TAU group will continue to receive their care as usual and be put on a waitlist. They will be offered the MBCT treatment after the completion of the study.

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy — A manualized 8-week MBCT group skills program with weekly sessions that each last 2 hours. The MBCT sessions combine elements of cognitive therapy with a mindful approach to thoughts and feelings, including a significant meditation component. The program is specifically tailored to a population that suffers from active depressive symptoms and chronic pain. The program also includes daily homework exercises.
  Arms: Treatment As Usual + Mindfulness Based Cognitive Therapy

SUMMARY:
The primary aim of this study is to test the feasibility and efficacy of Mindfulness Based Cognitive Therapy (MBCT) training for the treatment of depressive symptoms in patients with chronic pain. The study also aims to elucidate the mechanisms underlying MBCT on a psychological and neurobiological level. For this purpose the study subjects will fill out several psychological questionnaires related to mindfulness, depression and chronic pain. Moreover this study involves optional fMRI scans of the brain and blood measures before and after the intervention.

Main hypotheses:

1. The MBCT training will be a feasible intervention in patients with chronic pain and co-morbid depression as defined by no occurrence of serious adverse events related to the intervention and a retention rate of more than 70% in the subjects assigned to the MBCT arm.
2. Patients who have completed the MBCT training will demonstrate a significant decrease in depressive symptoms as measured on the Quick Inventory of Depressive Symptomatology - Clinician rated (QIDS-C16), and the Hamilton Rating Scale for Depression (HRSD17) (QIDS-C/HRDS) severity scale for depressive symptoms (the primary outcome measure), compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* The presence of Chronic Pain, which has persisted for at least 3 months.
* Meets criteria of Major Depressive Disorder, Dysthymic Disorder or Depressive disorder NOS as defined by DSM-IV criteria.
* Have a minimum score of depressive symptoms of > 10 as rated on the QIDS-C, administered during the screen.
* Able to provide written informed consent.
* Adults 18 years or older
* English-language literacy.

Exclusion Criteria:

* Serious suicide or homicide risk, as assessed by evaluating clinician.
* Severe and unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological or hematological disease for which hospitalization is likely to be required within the next half year.
* The following DSM-IV disorders: any bipolar disorder (current or past), current psychotic symptoms, or a primary psychotic disorder (current or past). Entry of patients with anxiety disorder will be permitted if the depressive disorder is judged to be the predominant disorder, in order to increase accrual of a clinically relevant sample.
* Active diagnosis of substance abuse or dependence disorders within the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline on the combined Quick Inventory of Depressive Symptomatology-clinician rated and the Hamilton Rating Scale for Depression (QIDS-C16/HRDS17), at week 8. | week 8

SECONDARY OUTCOMES:
Response according to the Beck Anxiety Inventory, 21 items (BAI). | Baseline, week 8, 6 months, 12 months
Response according to Short Form Health Survey, 36 items (SF-36). | Baseline, week 8, 6 months, 12 months
Response according to Brief Pain Inventory (BPI-sf). | Baseline, week 4, week 8, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Ashih, MD, PhD, Principal Investigator — Massachusetts General Hospital; Marasha De Jong, MD, Principal Investigator — Masachusetts General Hospital
Locations (1):
- MGH Depression Clinical and Research Program, Boston, Massachusetts, United States

REFERENCES:
- [Background] Teasdale JD, Segal ZV, Williams JM, Ridgeway VA, Soulsby JM, Lau MA. Prevention of relapse/recurrence in major depression by mindfulness-based cognitive therapy. J Consult Clin Psychol. 2000 Aug;68(4):615-23. doi: 10.1037//0022-006x.68.4.615. PMID 10965637
- [Background] Veehof MM, Oskam MJ, Schreurs KMG, Bohlmeijer ET. Acceptance-based interventions for the treatment of chronic pain: a systematic review and meta-analysis. Pain. 2011 Mar;152(3):533-542. doi: 10.1016/j.pain.2010.11.002. Epub 2011 Jan 19. PMID 21251756
- [Derived] de Jong M, Peeters F, Gard T, Ashih H, Doorley J, Walker R, Rhoades L, Kulich RJ, Kueppenbender KD, Alpert JE, Hoge EA, Britton WB, Lazar SW, Fava M, Mischoulon D. A Randomized Controlled Pilot Study on Mindfulness-Based Cognitive Therapy for Unipolar Depression in Patients With Chronic Pain. J Clin Psychiatry. 2018 Jan/Feb;79(1):15m10160. doi: 10.4088/JCP.15m10160. PMID 28252881
- See also: Depression Clinical and Research Program — http://www.massgeneral.org/psychiatry/services/treatmentprograms.aspx?id=1156